CLINICAL TRIAL: NCT01583543
Title: Phase II Study of the PARP Inhibitor, Olaparib, in Adult Patients With Recurrent/Metastatic Ewing's Sarcoma Following Failure of Prior Chemotherapy
Brief Title: Olaparib in Adults With Recurrent/Metastatic Ewing's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Edwin Choy, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-470
Record Dates: First submitted 2012-04-18; First posted 2012-04-24 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Ewing's Sarcoma
Keywords: Recurrent; Metastatic
MeSH Terms: conditions — Sarcoma, Ewing; Recurrence; Neoplasm Metastasis | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Olaparib (Experimental): 400mg PO BID Continuous
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — 400mg PO BID Continuous
  Other Names: AZD 2281

SUMMARY:
This research study is a Phase II clinical trial to test the efficacy of Olaparib in adult participants with recurrent/metastatic Ewing's Sarcoma following failure of prior chemotherapy.

DETAILED DESCRIPTION:
Primary Objectives Evaluate the objective response rate of olaparib in adult patients with recurrent and/or metastatic Ewing's sarcoma following failure of conventional chemotherapy.

Secondary Objectives To evaluate the progression-free survival, overall survival, and safety of olaparib in this patient population (ie Number of Participants With Adverse Events). As an exploratory objective, the investigators will evaluate (in subjects who agree to an optional biopsy) differences in pre- and post-treatment tumor DNA alterations and differences in levels of protein and RNA expression related to PARP inhibition.

Study Design Potential subjects who discuss and sign the informed consent form will undergo screening studies. Eligible patients will administer olaparib and obtain restaging imaging studies after 6 and 12 weeks on study, and then every 8 weeks thereafter. Participants will remain on study drug until disease progression, onset of unacceptable toxicities, or subject withdraws consent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Ewing's sarcoma
* Normal organ and bone marrow function
* Life expectancy of at least 16 weeks
* Not pregnant or breastfeeding
* Willing and able to comply with the protocol for the duration of the study
* Presence of measurable disease

Exclusion Criteria:

* Involvement in the planning and/or conduct of ths study
* Previous enrollment in the present study
* Participation in another clinical study with an investigational product during the 21 days prior to first dose of study drug
* Previous exposure to any PARP inhibitor
* Receiving systemic chemotherapy or radiotherapy within 2 weeks of beginning study treatment
* Receiving prohibited classes of inhibitors of CYP3A4
* Persistent clinically significant toxicities caused by previous cancer therapy
* Known myelodysplastic syndrome or acute myeloid leukemia
* Symptomatic, uncontrolled brain metastases
* Major surgery within 14 days of starting study treatment
* Considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disorder or active, uncontrolled infection
* Unable to swallow orally administered medication or with gastrointestinal disorders likely to interfere with absorption of the study medication
* Known to be serologically positive for HIV and receiving antiretroviral therapy
* Known active Hepatitis B or C
* Known hypersensitivity to olaparib or any of the excipients of the product
* Uncontrolled seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Choy, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Choy E, Butrynski JE, Harmon DC, Morgan JA, George S, Wagner AJ, D'Adamo D, Cote GM, Flamand Y, Benes CH, Haber DA, Baselga JM, Demetri GD. Phase II study of olaparib in patients with refractory Ewing sarcoma following failure of standard chemotherapy. BMC Cancer. 2014 Nov 5;14:813. doi: 10.1186/1471-2407-14-813. PMID 25374341

RESULTS

PARTICIPANT FLOW:
Groups:
- Olaparib: Patients with metastatic Ewing sarcoma who had previously received at least one line of chemotherapy were enrolled.
Period: Overall Study
Arm/Group | Olaparib
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Olaparib
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (15.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate of Olaparib
Description: Number of participants with objective response rate as defined as PR+CR as determined by RECIST vs. 1.1.
  Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib
Number analyzed (Participants) | 12
Participants | 0

2. Secondary Outcome: Progression-Free Survival
Description: Number of patients with progression free survival after two years from starting the trial.
Time Frame: Two years
Measure: Count of Participants; unit: Participants
Groups:
- Olaparib: This group of patients with metastatic Ewing sarcoma received single agent olaparib.
Arm/Group | Olaparib
Number analyzed (Participants) | 12
Participants | 0

3. Secondary Outcome: Overall Survival
Description: Number of patients survived for 2 years after enrolling onto this study.
Time Frame: Two years
Measure: Count of Participants; unit: Participants
Groups:
- Olaparib: This group of patients with metastatic Ewing sarcoma received single agent olaparib therapy.
Arm/Group | Olaparib
Number analyzed (Participants) | 12
Participants | 1

4. Secondary Outcome: Number of Participants Experiencing a Grade 3 or 4 Clinically Significant and Related Adverse Event
Description: Adverse events were graded according to CTCAE v.4 (Common Terminology Criteria for Adverse Events). Events are graded on a scale of 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, 5 = fatal. Only events that are clinically significant and which the treating investigator considers to be related to administration of olaparib are counted for this outcome measure.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib
Number analyzed (Participants) | 12
Participants | 4

ADVERSE EVENTS:
Time Frame: From initiation of study drug, throughout the study, and for 30 days after the last dose of study drug.
Groups:
- Olaparib: 400 mg PO BID Continuous Olaparib
Arm/Group | Olaparib
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olaparib (N=12)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Death (General disorders) | 2 — due to progressive disease
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olaparib (N=12)
Anemia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Sensitive teeth (Gastrointestinal disorders) | 1
Edema - limbs (General disorders) | 2
Fatigue (General disorders) | 3
Fever (General disorders) | 2
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 4
Allergies (Immune system disorders) | 1
Pneumonia (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Infection, other (Infections and infestations) | 2
Food poisoning (Injury, poisoning and procedural complications) | 1
Lymphopenia (Investigations) | 1
Thrombocytopenia (Investigations) | 2
Urinary hesitancy (Renal and urinary disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Polydipsia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Pain - other (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
headache (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Perinea/ Genital numbness (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Cellulitis (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 1
Lymphedema (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No